CLINICAL TRIAL: NCT00856765
Title: Randomized Comparison of Drug Eluting Balloon/Bare Metal Stent Versus Drug Eluting Stent Versus Bare Metal Stent for the Treatment of Patients With Acute ST-elevation Myocardial Infarction
Brief Title: Drug-eluting Balloon in Acute Myocardial Infarction
Acronym: DEB-AMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Prof. Pieter Stella, PHD.MD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METC 08-255
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Thrombosis; Acute Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Thrombosis | interventions — Magic; Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Drug eluting balloon followed immediately by implantation of bare metal stent
  Interventions: Device: Drug eluting balloon; Device: Bare metal stent
- 2 (Active Comparator): Drug eluting stent
  Interventions: Device: Drug eluting stent
- 3 (Active Comparator): Bare metal stent
  Interventions: Device: Bare metal stent

INTERVENTIONS:
Device: Drug eluting balloon — Percutaneous transluminal coronary balloon angioplasty catheter eluting paclitaxel
  Other Names: Dior (EuroCor)
  Arms: 1
Device: Bare metal stent — Bare metal stent
  Other Names: Magic (EuroCor)
  Arms: 1; 3
Device: Drug eluting stent — Paclitaxel eluting stent
  Other Names: Taxus Liberté (Boston scientific)
  Arms: 2

SUMMARY:
The investigators hypothesize that patients with Acute ST Elevation Myocardial Infarction may benefit from primary angioplasty with use of a drug eluting balloon/bare metal stent combination without impairing the process of normal vascular healing and endothelial function.

The goals of this study are:

1. To compare 6-month angiographic outcome after primary angioplasty using drug eluting balloon/bare metal stent combination versus drug eluting stent versus bare metal stent.
2. To compare stent apposition and stent endothelialization after primary angioplasty using drug eluting balloon/bare metal stent versus drug eluting stent versus bare metal stent.
3. To compare coronary endothelial function after primary angioplasty using drug eluting balloon/bare metal stent versus drug eluting stent versus bare metal stent.

ELIGIBILITY:
Inclusion Criteria:

* STEMI within 12 hours of onset of complaints
* Candidate for primary PCI with stent-implantation
* Successful thrombus aspiration defined by no angiographic signs of thrombus a the site of plaque rupture and TIMI flow more or equal 1

Exclusion Criteria:

* Unable to give written informed consent
* Diabetes and Type C- coronary lesion
* Previous PCI or CABG of infarct related vessel
* Left main stenosis more than 50%.
* Triple vessel disease with stenosis more than 50% in 3 epicardial coronary arteries
* Target vessel reference diameter less than 2.5 and more than 4.0 mm
* Target lesion length more than 25 mm
* Intolerance for aspirin or clopidogrel
* Life expectancy less than 12 months
* Women with child bearing potential

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Angiographic in-segment late lumen loss (expressed in millimeters) as determined by quantitative coronary analysis (QCA) | 6 months

SECONDARY OUTCOMES:
Binary restenosis using QCA | 6 months
stent malapposition and re-endothelialization assessed by Optical Coherence Tomography (OCY) | 6 months
coronary endothelial dysfunction after acetylcholine infusion | 6 months
Clinical outcomes (death, myocardial infarction, repeated revascularization procedures) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Stella, MD, Principal Investigator — UMC Utrecht
Locations (2):
- University of Modena, Department of Cardiology, Modena, Italy
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Belkacemi A, Agostoni P, Nathoe HM, Voskuil M, Shao C, Van Belle E, Wildbergh T, Politi L, Doevendans PA, Sangiorgi GM, Stella PR. First results of the DEB-AMI (drug eluting balloon in acute ST-segment elevation myocardial infarction) trial: a multicenter randomized comparison of drug-eluting balloon plus bare-metal stent versus bare-metal stent versus drug-eluting stent in primary percutaneous coronary intervention with 6-month angiographic, intravascular, functional, and clinical outcomes. J Am Coll Cardiol. 2012 Jun 19;59(25):2327-37. doi: 10.1016/j.jacc.2012.02.027. Epub 2012 Apr 11. PMID 22503057